CLINICAL TRIAL: NCT06909175
Title: Comparing Transesophageal Echocardiography and Trans Abdominal Doppler for Portal Vein Assessment in Living Donor Liver Transplantation
Brief Title: Comparing Portal Vein Assessment by Intraoperative Doppler and Transesophageal Echocardiography
Status: Completed | Type: Observational
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Principal Investigator, Gaurav Sindwani, Associate Professor, Institute of Liver and Biliary Sciences, India
Other Study IDs: ILBSindia5
Record Dates: First submitted 2025-03-27; First posted 2025-04-03 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Chronic Liver Disease
MeSH Terms: interventions — Echocardiography, Transesophageal

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Transesophageal echocardiography — Portal vein velocities were measured using TEE and intraoperative doppler in patients undergoing living donor liver transplantation

SUMMARY:
Liver transplantation is usually associated with hemodynamic instability. TEE allows for a real time monitoring of cardiac structures and has become a standard of care for liver transplant patients. Society of cardiovascular anaesthesia and American society of anaesthesiologists recommends use of TEE in non-cardiac surgery patients with hemodynamic instability. Also, society for advancement of transplant anaesthesia (SATA) has suggested that TEE usage in cases of liver transplant is safe, effective and improves outcomes. TEE can also provide vital information relating to non-cardiac structures including liver, spleen, kidneys, portal vein, hepatic vein and other major vessels. As of now standard protocol is to do the transabdominal doppler for the assessment of portal vein after the liver graft implantation. Hence, the aim of our study is to compare the transesophageal echocardiography and transabdominal Doppler for assessing portal vein in living donor liver transplantation.

DETAILED DESCRIPTION:
Data from all patients who underwent live donor liver transplant surgery at Institute of Liver and Biliary Sciences, New Delhi and in whom TEE probe was inserted will be collected and analysed.

ELIGIBILITY:
Inclusion Criteria:

* All patients who have undergone Live donor liver transplant, Age > 18 years

Exclusion Criteria:

* Required data is not available

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Chronic liver disease
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2025-04-05 (Actual); Primary Completion 2025-05-05 (Actual); Study Completion 2025-06-05 (Actual)

PRIMARY OUTCOMES:
To compare the portal vein flow velocity using transesophageal echocardiography and transabdominal Doppler during live donor liver transplant surgery. | intraoperative period

SECONDARY OUTCOMES:
any TEE related complication | intraoperative period

CONTACTS AND LOCATIONS:
Overall Officials: Gaurav Sindwani, MD, Principal Investigator — Institute of Liver and Biliary Sciences
Locations (1):
- ILBS, Delhi, India

IPD SHARING:
Plan to Share IPD: No